CLINICAL TRIAL: NCT05018962
Title: Recurrent Stenoses in Arteriovenous Fistula (AVF) for Dialysis Access: CuttIng ballooN angioplaSTy Combined wITh Paclitaxel drUg coaTed Balloon Angioplasty, an observatIONal Clinical Study
Acronym: INSTITUTION
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Singapore General Hospital (Other)
Collaborators: Boston Scientific Corporation (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2017/2046
Record Dates: First submitted 2021-08-22; First posted 2021-08-24 (Actual); Last update posted 2021-08-24 (Actual); Status verified 2021-08

CONDITIONS: Dialysis Access Malfunction
Keywords: Paclitaxel coated balloon; Cutting balloon; Recurrent stenosis
MeSH Terms: conditions — Constriction, Pathologic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (1):
- Cutting balloon followed by paclitaxel coated balloon (Experimental)
  Interventions: Device: Cutting balloon followed by paclitaxel coated balloon

INTERVENTIONS:
Device: Cutting balloon followed by paclitaxel coated balloon — Cutting balloon followed by paclitaxel coated balloon

SUMMARY:
To determine if cutting balloon angioplasty combined with DEB angioplasty provides a higher primary patency after treatment of recurrent stenoses compared with cutting balloon angioplasty or angioplasty using DEB alone in the venous outflow AVFs. For cutting balloon angioplasty in venous stenosis, the primary patency after 12 months is 55-60% (9,16) and in recurrent stenoses up to 48%(10).

We hypothesise that DEB angioplasty after cutting balloon angioplasty leads to improved primary patency at 12 months.

ELIGIBILITY:
Inclusion Criteria:

* Recurrent stenoses (within 1 year after angioplasty) in the venous outflow of AVFs for dialysis access (> 0.5cm from AV anastomosis up to cephalic arch)
* Successful guidewire crossing of target lesion
* ≥ 21 years old
* Informed and valid consent given.
* Patient willing and able to return for follow up .

Exclusion Criteria:

1. Thrombosed AVFs or occlusions in the access circuit
2. Significant cephalic arch (central perpendicular portion of the cephalic vein) or central vein stenoses.
3. > 3 stenosed segments (lesions are considered separate if they are separated by at least 2 cm normal vessel.)
4. Only potential target lesion located in cephalic arch, central veins or anastomotic lesions.
5. Only de novo stenoses identifiable as target lesion.
6. Target lesion resistant to cutting balloon angioplasty (>30% residual stenosis with incomplete effacement of the lesion during cutting balloon angioplasty)
7. Target lesion not treatable with the available sizes of cutting balloon (4-7mm) and drug eluting balloon (up to 8mm) so native reference vessel <3 mm or need for DEB balloon >8mm.
8. Lesion in excess of 8 cm
9. Unable to take dual antiplatelet therapy for 1 month and/or aspirin for 6 months
10. Coagulopathy (PT or PTT >1.5 times the median of normal range) or thrombocytopenia (platelet count <50,000 /μL) that cannot be managed adequately with periprocedural transfusion.
11. Patient on Warfarin.
12. Known allergy to iodinated contrast that cannot be managed adequately with pre-procedure medication.
13. Allergy / contraindication to dual anti-platelet therapy (aspirin and clopidogrel or ticlopidine) or paclitaxel.
14. Acute infection over proposed puncture site.
15. Women who are breastfeeding, pregnant or planning on becoming pregnant during study.
16. Participant with medical conditions, which in the opinion of the investigator may cause non-compliance with protocol.
17. Currently participating in an investigational drug, biologic or device trial that may have an impact on the dialysis access or previous enrolment in this study.

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 44 (Actual)
Dates: Start 2017-09-08 (Actual); Primary Completion 2019-04-15 (Actual); Study Completion 2020-03-18 (Actual)

PRIMARY OUTCOMES:
Target lesion primary patency | 1 year
  Target lesion primary patency

SECONDARY OUTCOMES:
Circuit primary patency | 1 year
  Circuit primary patency
Target lesion primary assisted patency | 1 year

CONTACTS AND LOCATIONS:
Locations (1):
- Singapore General Hospital, Singapore, Singapore

IPD SHARING:
Plan to Share IPD: No